CLINICAL TRIAL: NCT03771937
Title: The Effect of Education and Telephone Follow-up Intervention Based on the Roy Adaptation Model After Myocardial Infarction: a Randomized Controlled Trial
Brief Title: The Effect of Education and Telephone Follow-up Intervention Based on the Roy Adaptation Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Selma Turan, Nursing Faculty, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0001
Record Dates: First submitted 2018-12-05; First posted 2018-12-11 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Myocardial Infarction
Keywords: lifestyle change; telephone follow-up; Roy Adaptation Model
MeSH Terms: conditions — Myocardial Infarction | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinding was provided that included inclusion criteria and agreement to participate in the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group received a telephone follow-up intervention, which consisted of a pre-discharge education program and three telephone follow-up sessions based on the RAM.
  Interventions: Other: Education and telephone follow-up intervention
- Control group (No Intervention): the control group received routine care.

INTERVENTIONS:
Other: Education and telephone follow-up intervention — A telephone follow up and a pre-discharge education
  Arms: Intervention

SUMMARY:
In this parallel randomized controlled trial (n = 33/group), the control group received routine care, while the intervention group received a telephone follow-up intervention, which consisted of a pre-discharge education program and three telephone follow-up sessions based on the Roy Adaptation Model.

DETAILED DESCRIPTION:
Objective: To evaluate the effect of education and telephone follow-up intervention based on the Roy Adaptation Model (RAM) for improving MI patients' self-efficacy, quality of life and lifestyle adaptation.

Methods: In this parallel randomized controlled trial (n = 33/group), the control group received routine care, while the intervention group received a telephone follow-up intervention, which consisted of a pre-discharge education program and three telephone follow-up sessions based on the RAM. Data were collected before discharge, and in the 12th week after discharge included quality of life, coping adaptation process, self-efficacy and lifestyle changes.

ELIGIBILITY:
Inclusion Criteria:

1. Participants were adults aged ≥30 years and had been admitted to the hospital with a diagnosis of MI (which must be supported by ECG and an increase in biomarkers).
2. were clinically stable
3. willing to participate
4. able to understand and write Turkish
5. able to receive telephone calls or fill in questionnaires.
6. able to come to the hospital for checkups. Exclusion Criteria:Patients were excluded from the study if according to medical file records they had chronic renal failure, cancer, heart failure, severe aortic stenosis, if they were planned for surgical treatment or had chronic cognitive and psychiatric disease, if they had problems with hearing and speaking on the phone, or if they had mobility restriction.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-04-03 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
General Self-Efficacy Scale | 12 week
  The self-efficacy levels of the patients were measured by the General Self-Efficacy Scale (GSES). The GSES contains 10 items and each item score ranges from 0 to 5. Cronbach's α of the GSES was 0.83. The highest and lowest possible score is between 10-40. High score indicates that the individual perceives high self-efficacy.
Coping and Adaptation scale | 12 week
  To evaluate the coping and adaptation processes, the Coping and Adaptation (CAPS) scale was used. The CAPS was developed by Callista Roy. The Turkish validity and reliability study of the scale was conducted by Çatal and Dicle (2015), and the Cronbach alpha value was 0.82 for the total scale. The highest and lowest possible score is between 47-188. Higher scores indicate better use of effective coping methods.
Myocardial Infarction Dimensional Assessment Scale | 12 week
  To evaluate the quality of life after the disease, the Myocardial Infarction Dimensional Assessment Scale (MIDAS) was used. This was developed by Thompson et al. in 2002. The Cronbach alpha values of the scale were found in seven dimensions, and ranged from 0.74 to 0.95, showing it to be a useful and highly reliable tool. The validity and reliability study of the scale was made by Yilmaz et al. Cronbach alpha values ranged from 0.79 to 0.90. The 10 highest and lowest possible score is between 0-100, with 0 indicating the best health condition, and 100 indicating the worst health condition.

CONTACTS AND LOCATIONS:
Overall Officials: Selma Turan Kavradım, PhD, Principal Investigator — Akdeniz University Nursing Faculty; Zeynep Canlı ÖZER, Professor, Study Director — Akdeniz University Nursing Faculty

IPD SHARING:
Plan to Share IPD: No
The investigators plan to send the results to an international journal and all results can be obtained after publication.